CLINICAL TRIAL: NCT02095678
Title: Assessment of Novel MRI Quantification Free Breathing Technique in Evaluation of Liver Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE3213
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma; Liver Cell Carcinoma, Adult; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HCC or metastatic Liver Lesions (Experimental): Patients with HCC or metastatic liver lesions who are refered to the abdominal imaging and biopsy clinic will have a liver biopsy performed. 3-5 days after a clinical MRI indicating a cancerous lesion, patients will return for the free-breathing MRI and a liver biopsy. These images will be compared to the clinical MRI and to images of the benign lesions.
  Interventions: Procedure: liver biopsy; Device: free-breathing MRI
- Benign Liver Lesion (Active Comparator): Patients with benign liver lesions will be referred to the study team. 3-5 days after a clinical MRI an experimental, free-breathing MRI will be performed on these patients. The results will be compared to their clinical MRI images and to images of HCC or metastatic lesions
  Interventions: Device: free-breathing MRI

INTERVENTIONS:
Procedure: liver biopsy — patients with HCC or metastatic lesions will have a liver biopsy performed after the experimental MRI. This biopsy will be examined to confirm the imaging results
  Arms: HCC or metastatic Liver Lesions
Device: free-breathing MRI — All patients will be asked to come in for an MRI scan using techniques developed which minimize the time a patient has to hold their breath to image the liver to <8 seconds and validate quantifiable techniques which improve liver image quality
  Other Names: experimental MRI

SUMMARY:
The primary objective of this study is to develop and validate simultaneous free-breathing 4D fat and water quantification and quantitative dynamic contrast enhanced perfusion in the liver. Secondary aims include developing and validating free breathing quantification of relaxation parameters T1 and T2, and developing and validating a minimal breath-hold (< 8 s) high quality diffusion exam using highly accelerated steady state diffusion imaging sequences. Investigators aim to scan 100 subjects receiving liver biopsies as a part of their standard care and another 70 subjects with known benign lesions. The study is greater than minimal risk.

DETAILED DESCRIPTION:
The investigators hypothesize that a quantitative and near free-breathing MRI approach with Hepatocellular carcinoma (HCC) patients will lead to improved tissue characterization, resulting in fewer ambiguous readings and thus fewer biopsies. As each component of the proposed methodology has been experimentally validated in the investigators preliminary work, the next appropriate step would be to evaluate the clinical feasibility of the exam. The investigators goal is to test the ability of quantitative MRI techniques to provide high quality images of the liver and to differentiate liver lesions from one another in a time frame shorter than a current clinical exam.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to getting contrast enhanced MRI examinations.
* GFR ≥ 40.

Exclusion Criteria:

* Patients with ferromagnetic or otherwise non-MRI compatible aneurysm clips.
* The presence of an implanted pacemaker or implanted defibrillator device
* Patients with contraindications for MRI due to embedded foreign metallic objects. Bullets, shrapnel, metalwork fragments, or other metallic material adds unnecessary risk to the patient.
* Pregnancy. Regular clinical practice already excludes pregnant patients from gadolinium contrast due to unknown effects on the fetus. The current clinical practice will be applied - patients will be verbally screened and asked if they think they could be pregnant. If the answer is yes, then the patient will be excluded from the study. If the patient is uncertain about the pregnancy status, she will be given an option to undergo a pregnancy test or not participate in the study altogether. Patients who self report that they are not pregnant will be allowed to participate in the study. This procedure is based on current department policy guidelines.
* Implanted medical device not described above that is not MRI-compatible;
* Known history of claustrophobia;
* Known history of allergic reaction to Magnetic Resonance contrast material;
* Late stage renal failure with estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73 m2 based on patient's serum creatinine due to the significantly increased risk of nephrogenic systemic fibrosis (NSF). ('Past' 3 months timeframe will be used to calculate the eGRF).
* Minors will be excluded.
* Prisoners and members of other vulnerable populations will be excluded from this study. The subject selection population will not regularly include prisoners and other vulnerable population members as these populations will not provide any additional unique information to or uniquely benefit from the study. Non-english speaking population will be excluded from the study due to lack of sufficient resources to pay for translator and interpreter services.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-12-01; Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gulani, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Pahwa S, Liu H, Chen Y, Dastmalchian S, O'Connor G, Lu Z, Badve C, Yu A, Wright K, Chalian H, Rao S, Fu C, Vallines I, Griswold M, Seiberlich N, Zeng M, Gulani V. Quantitative perfusion imaging of neoplastic liver lesions: A multi-institution study. Sci Rep. 2018 Mar 21;8(1):4990. doi: 10.1038/s41598-018-20726-1. PMID 29563601

RESULTS

PARTICIPANT FLOW:
Groups:
- Dynamic Contrast Enhanced MRI: Patients with HCC or metastatic liver lesions who are refered to the abdominal imaging and biopsy clinic will have a liver biopsy performed. 3-5 days after a clinical MRI indicating a cancerous lesion, patients will return for the free-breathing MRI and a liver biopsy. These images will be compared to the clinical MRI and to images of the benign lesions.
  liver biopsy: patients with HCC or metastatic lesions will have a liver biopsy performed after the experimental MRI. This biopsy will be examined to confirm the imaging results
  free-breathing MRI: All patients will be asked to come in for an MRI scan using techniques developed which minimize the time a patient has to hold their breath to image the liver to <8 seconds and validate quantifiable techniques which improve liver image quality
- Free-Breathing Quantification of Relaxation Parameters: Patients with benign liver lesions will be referred to the study team. 3-5 days after a clinical MRI an experimental, free-breathing MRI will be performed on these patients. The results will be compared to their clinical MRI images and to images of HCC or metastatic lesions
  free-breathing MRI: All patients will be asked to come in for an MRI scan using techniques developed which minimize the time a patient has to hold their breath to image the liver to <8 seconds and validate quantifiable techniques which improve liver image quality
Period: Overall Study
Arm/Group | Dynamic Contrast Enhanced MRI | Free-Breathing Quantification of Relaxation Parameters
Started | 34 | 18
Completed | 17 | 0
Not Completed | 17 | 18
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Omitted for Severe Image Artifacts or Patient Non-compliance | 11 | 12
Not completed — lesion impacted by previous treatment | 1 | 1
Not completed — No Confirmed Diagnosis | 0 | 3
Not completed — Malignant lesions not HCC nor Metastatic | 1 | 1
Not completed — No Visible Lesion or Pathological Finding | 4 | 0

BASELINE CHARACTERISTICS:
Population: Participants that had evaluable scans.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dynamic Contrast Enhanced MRI | Free-Breathing Quantification of Relaxation Parameters | Total
Number analyzed (Participants) | 34 | 18 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 13 | 31
  >=65 years | 16 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 22 | 13 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 18 | 52
Lesion type [Count of Participants; unit: Participants]
  HCC | 10 | 9 | 19
  Metastatic Cancer | 16 | 3 | 19
  Benign | 3 | 2 | 5
  No confirmed diagnosis, other malignant, or no visible lesion/path | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Arterial Fraction
Description: Dynamic Contrast Enhanced MRI data were used to calculate three quantitative perfusion properties using a dual input, single tissue compartment model of gadolinium based contrast agents in the liver in HCC, metastatic, and benign lesions.
  One of these quantitative perfusion properties is Mean Arterial fraction, which is the proportion of blood flow derived from hepatic artery.
Time Frame: 1 day, At time of Research MRI
Population: Evaluable participants (those who completed study with applicable lesions). Note - There were only sufficient number of participants to statistically compare HCC and Metastatic lesion groups due to the low number of benign lesions. No data are available for the "Free-breathing Quantification of Relaxation Parameters" for reasons listed in participant flow section - primarily relating to image blurring and artifacts.
Measure: Mean (Standard Deviation); unit: percentage of arterial fraction
Units Other Than Participants: Lesions
Groups:
- Dynamic Contrast Enhanced MRI - HCC Lesions; Dynamic Contrast Enhanced MRI - Metastatic Lesions; Dynamic Contrast Enhanced MRI - Benign Lesions: Patients with HCC or metastatic liver lesions who are refered to the abdominal imaging and biopsy clinic will have a liver biopsy performed. 3-5 days after a clinical MRI indicating a cancerous lesion, patients will return for the free-breathing MRI and a liver biopsy. These images will be compared to the clinical MRI and to images of the benign lesions.
  liver biopsy: patients with HCC or metastatic lesions will have a liver biopsy performed after the experimental MRI. This biopsy will be examined to confirm the imaging results free-breathing MRI: All patients will be asked to come in for an MRI scan using techniques developed which minimize the time a patient has to hold their breath to image the liver to <8 seconds and validate quantifiable techniques which improve liver image quality
Arm/Group | Dynamic Contrast Enhanced MRI - HCC Lesions | Dynamic Contrast Enhanced MRI - Metastatic Lesions | Dynamic Contrast Enhanced MRI - Benign Lesions
Number analyzed (Participants) | 5 | 10 | 2
Number analyzed (Lesions) | 13 | 46 | 3
percentage of arterial fraction | 79.8 (12.9) | 72.2 (20.4) | 73.6 (15.9)
Statistical Analysis 1: Comparison: Dynamic Contrast Enhanced MRI - HCC Lesions vs Dynamic Contrast Enhanced MRI - Metastatic Lesions; Test type: Other — Significance (alpha) set to 0.05; p = 0.211, t-test, 2 sided

2. Secondary Outcome: Free Breathing Quantification of Relaxation Parameters
Description: Quantified and validated relaxation parameters when creating T1 (spin-lattice) and T2 (spin-spin) weighted images
Time Frame: Up to 1 year
Population: Quality of images were poor and could not be used for analysis
Arm/Group | Dynamic Contrast Enhanced MRI | Free-Breathing Quantification of Relaxation Parameters
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Minimal Breathhold Time
Description: The minimum time (in seconds) a patient must hold their breath to produce quality liver images during an MRI. Developing and validating a minimal breath-hold (< 8 s) high quality diffusion exam using highly accelerated steady state diffusion imaging sequences.
Time Frame: 1 year
Population: Although the study team worked on the development of this technology as part of an NIH grant, this technology was not utilized as a part of this study so no data were collected.
Arm/Group | Dynamic Contrast Enhanced MRI | Free-Breathing Quantification of Relaxation Parameters
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Distribution Volume (DV)
Description: Dynamic Contrast Enhanced MRI data were used to calculate three quantitative perfusion properties using a dual input, single tissue compartment model of gadolinium based contrast agents in the liver in HCC, metastatic, and benign lesions.
  One of these quantitative perfusion properties is DV. DV corresponds to the volume of extracellular, extravascular space in a tissue which is a measure of the tissue cellularity
Time Frame: 1 day, At time of Research MRI
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of DV
Units Other Than Participants: Lesions
Arm/Group | Dynamic Contrast Enhanced MRI - HCC Lesions | Dynamic Contrast Enhanced MRI - Metastatic Lesions | Dynamic Contrast Enhanced MRI - Benign Lesions
Number analyzed (Participants) | 5 | 10 | 2
Number analyzed (Lesions) | 13 | 46 | 3
percentage of DV | 29.9 (13.0) | 53.8 (19.3) | 61.8 (20.9)
Statistical Analysis 1: Comparison: Dynamic Contrast Enhanced MRI - HCC Lesions vs Dynamic Contrast Enhanced MRI - Metastatic Lesions; Test type: Other — Significance (alpha) set to 0.05; p < 0.01, t-test, 2 sided

5. Primary Outcome: Mean Transit Time (MTT)
Description: Dynamic Contrast Enhanced MRI data were used to calculate three quantitative perfusion properties using a dual input, single tissue compartment model of gadolinium based contrast agents in the liver in HCC, metastatic, and benign lesions.
  One of these quantitative perfusion properties is MTT. MTT corresponds to the average time, in seconds, that red blood cells spend within a determinate volume of capillary circulation
Time Frame: 1 day, At time of Research MRI
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Lesions
Arm/Group | Dynamic Contrast Enhanced MRI - HCC Lesions | Dynamic Contrast Enhanced MRI - Metastatic Lesions | Dynamic Contrast Enhanced MRI - Benign Lesions
Number analyzed (Participants) | 5 | 10 | 2
Number analyzed (Lesions) | 13 | 46 | 3
seconds | 12.0 (3.1) | 44.6 (25.7) | 5.8 (2.0)
Statistical Analysis 1: Comparison: Dynamic Contrast Enhanced MRI - HCC Lesions vs Dynamic Contrast Enhanced MRI - Metastatic Lesions; Test type: Other — Significance (alpha) set to 0.05; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Within 48 hours of scan
Arm/Group | Dynamic Contrast Enhanced MRI | Free-Breathing Quantification of Relaxation Parameters
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/18
Other Adverse Events (participants affected / at risk) | 0/34 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynamic Contrast Enhanced MRI (N=34) | Free-Breathing Quantification of Relaxation Parameters (N=18)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Free breathing quantification of T1 and T2 was explored and initial tests were run as part of this study. However, free-breathing acquisition of data yielded substantial image blurring, making it impossible to accurately delineate and characterize lesions. Several technical improvements were implemented, but improved image quality was not achieved. Dynamic Contrast Enhanced MRI data from this study combined with data from a second institution were published in Nature Scientific Reports in 2018

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT02095678/Prot_SAP_002.pdf
  • Informed Consent Form (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02095678/ICF_001.pdf